CLINICAL TRIAL: NCT06024954
Title: Palliative Care Pain, Anxiety and Vital Inhaler Effect of Aromatherapy Applied to Patients and Music Effect on Parameters
Brief Title: Pain, Anxiety of Aromatherapy and Music Effect on
Acronym: Palliative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Duygu Akbas Uysal, Registered Nurse, Ege University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: EGE UNIVERSTY; DUYGU AKBAŞ UYSAL (Other: EGE UNIVERSTY)
Record Dates: First submitted 2023-07-11; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Cancer
Keywords: pallative care; aromatherapy; music therapy
MeSH Terms: conditions — Neoplasms | interventions — Aromatherapy; Music Therapy

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- music group (Experimental): The research is planned as a randomized controlled trial. The individuals in the research group are divided into four groups as music group, aromatherapy group, music and aromatherapy and control group. The relaxing music group will listen to specially composed "MusiCure®" compositions in soft rhythm, including melodies with harp, cello, strings and natural sound elements (eg rain, bird, forest sound). The patients in the experimental group will listen to the music with headphones for 20 minutes for three consecutive days.
  Before and at the end of the intervention, data collection tools [Patient Description Form, Vısual analog scale, facial anxiety scale , Distress Thermometer, Edmonton Symptom Scale] will record the characteristics of pain, anxiety and vital parameters.
  Interventions: Other: music therapy
- aromatherapy group (Experimental): Patients in the aromatherapy group use 5% lavender oil with a diffuser for 15-20 minutes in accordance with the "Aromatherapy-Clinical Guideline For Midwives. NHS".
  Trust 1-15) has been applied. The diffuser was placed 30 cm from the participants and five (5) drops of essential lavender oil were placed on the filter paper. Within 10-15 minutes after the completion of the inhalation, data collection forms were applied again, and pain, anxiety, blood pressure, pulse and respiratory rate were evaluated.
  Interventions: Other: aromatherapy
- aromatherapy and music group (Experimental): Inpatients in the palliative care service will be given music with headphones for three consecutive days with the effect of aromatherapy inhaler. Within 10-15 minutes after the completion of the inhalation, data collection forms will be applied again and pain, anxiety, blood pressure, pulse and respiratory rate will be evaluated.
  Interventions: Other: aromatherapy and music therapy
- control group (No Intervention): Participants were not interfered with.

INTERVENTIONS:
Other: aromatherapy — Patients in the aromatherapy group use 5% lavender oil with a diffuser for 15-20 minutes in accordance with the "Aromatherapy-Clinical Guideline For Midwives. NHS".
  Trust 1-15) has been applied. The diffuser was placed 30 cm from the participants and five (5) drops of essential lavender oil were placed on the filter paper. Within 10-15 minutes after the completion of the inhalation, data collection forms were applied again, and pain, anxiety, blood pressure, pulse and respiratory rate were evaluated.
  Other Names: aromatherapy inhaler.
  Arms: aromatherapy group
Other: music therapy — The relaxing music group listened to specially composed "MusiCure®" compositions in soft rhythm, including melodies with harp, cello, strings and sound elements from nature (eg rain, bird, forest sound). Listened with headphones for 20 minutes.
  Arms: music group
Other: aromatherapy and music therapy — Inpatients will be given music with a loudspeaker with the effect of aromatherapy inhaler for three consecutive days. Within 10-15 minutes after the completion of the inhalation, data collection forms will be applied again, pain, anxiety, blood pressure, pulse, respiratory rate were evaluated.
  Arms: aromatherapy and music group

SUMMARY:
The research is planned as a randomized controlled trial. The main question[s] it aims to answer are:

[question 1]: Does the inhaler effect of music and aromatherapy applied to palliative care patients have an effect on pain, anxiety and vital signs?

The individuals in the research group are divided into four groups as music group, aromatherapy group, music and aromatherapy and control group. .

Before and at the end of the intervention, data collection tools [Patient Description Form, Visual analog scale,face anxiety scale, Distress Thermometer, Edmonton Symptom Scale] will record the characteristics of pain, anxiety and vital parameters.

Patient Identification Form: It is a questionnaire that includes sociodemographic characteristics (gender, age, educational status, income status, employment status and occupation) and questions about the disease, created by the researchers by scanning the literature.

DETAILED DESCRIPTION:
The relaxing music group listened to specially composed "MusiCure®" compositions in soft rhythm, including melodies with harp, cello, strings and sound elements from nature (eg rain, bird, forest sound).The patients in the experimental group listened to music with headphones for 20 minutes for three consecutive days.Pain, anxiety and vital parameters were recorded with data collection tools [Patient Description Form, VAS, FAS, Distress Thermometer, Edmonton Symptom Scale] before and at the end of the intervention.For the patients in the aromatherapy group, use 5% lavender oil with a diffuser for 15-20 minutes.

has been applied.The diffuser was placed 30 cm from the participants and five (5) drops of essential lavender oil were placed on the filter paper. Within 10-15 minutes after the completion of the inhalation, data collection forms were applied again and pain, anxiety, blood pressure, pulse and respiratory rate were evaluated.The patients hospitalized in the palliative care service were given music with a loudspeaker for three consecutive days with the effect of aromatherapy inhaler.

Within 10-15 minutes after the completion of the inhalation, data collection forms were applied again and pain, anxiety, blood pressure, pulse and respiratory rate were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* who volunteered to participate in the research,
* 18 years and older,
* No hearing problem
* Doesn't have any problems with smelling healthy,
* No communication and speech problems

Exclusion Criteria:

* with a diagnosis of psychiatric illness,
* Allergic to lavender, perfumes or cosmetics,
* Having asthma and chronic obstructive pulmonary disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | three consecutive days after the start of application
  The Visual Analog Scale (VAS) used for the assessment of pain is used to digitize some values that cannot be measured numerically. Two end definitions of the parameter to be evaluated are written at both ends of a 10 cm or 100 mm line, and the patient is asked to indicate where on this line their situation is appropriate by drawing a line or by placing a dot or pointing.
Facial Anxiety Scale (FAS) | three consecutive days after the start of application
  The Facial Anxiety Scale is a measurement tool in which patients report their anxiety levels. The scale consists of five face shapes with the size of 11 × 42 cm. While the facial expression on the far left indicates the absence of anxiety, the level of anxiety increases towards the right (scored between 0-5). A score of three or more on the Facial Anxiety Scale indicates that the anxiety level is moderate or high.
Distress Thermometer | three consecutive days after the start of application
  Distress Thermometer The Thermometer with Distress Thermometer is a likert-type scale with scores from 0 (no stress) to 10 (extreme stress).the class of the values in the degree is indicated as points
Edmonton Symptom Diagnostic Scale((ESAS) | three consecutive days after the start of application
  The patient is asked to match his symptoms with a number that he thinks is most suitable for him from the numbers from 0 to 10. The number 0 indicates no symptoms, the number 10 indicates that the symptom is very severe.All of the items on the ESAS have a value of 0-10 points
vital parameters | three consecutive days after the start of application
  blood pressure measurement, pulse, respiratory rate will be measured.120-129/80-84 mmHg is normal, 130-139/85-89 mmHg( millimeters of mercury (mmHg) ) is called high normal blood pressure.Respirations per minute in a healthy adult person 12-20.(12-20 breaths per minute)It is normal for adults and healthy people to have a heart rate in the range of 60-100 beats per minute.Heart rate (or pulse rate)(heart per minute (beats per minute, or bpm)(60 to 100 bpm);

CONTACTS AND LOCATIONS:
Overall Officials: DUYGU AKBAŞ UYSAL, Principal Investigator — PHD.candidate
Locations (1):
- EGE, Izmir, İ̇zmi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akbas Uysal D, Senuzun Aykar F, Uyar M. The effects of aromatherapy and music on pain, anxiety, and stress levels in palliative care patients. Support Care Cancer. 2024 Sep 4;32(10):632. doi: 10.1007/s00520-024-08837-0. PMID 39230757